CLINICAL TRIAL: NCT00212875
Title: An Open-Label, Randomized, Multicenter Study of the Initiation of Four Dosing Regimens of PROCRIT (Epoetin Alfa) for the Treatment of Anemia of Chronic Kidney Disease (CKD). Protocol Addendum: Due to Space Constraints, See Detailed Description for Full Title of Addendum.
Brief Title: A Study of Four Dosing Regimens of PROCRIT (Epoetin Alfa) in Patients With Chronic Kidney Disease. Protocol Addendum: Extension Study of Maintenance Therapy of PROCRIT (Epoetin Alfa) in Patients With Chronic Kidney Disease.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Centocor Ortho Biotech Services, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR003397; NCT00246311 (obsolete NCT alias)
Record Dates: First submitted 2005-09-16; First posted 2005-09-21 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2010-03

CONDITIONS: Chronic Kidney Disease; Anemia
Keywords: Chronic Kidney disease; anemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The primary objective of this study is to compare the change in hemoglobin (Hb) from study start to the end of the study between the every 2 week and the every 4 week dosing regimens in patients with anemia of chronic kidney disease (CKD) initiated on PROCRIT (epoetin alfa). Protocol Addendum: The primary objective of the open-label extension portion of this study is to evaluate if epoetin alfa 40,000 Units given under the skin every six weeks, can maintain hemoglobin within the range of 11-12 g/dL in patients with anemia of CKD.

DETAILED DESCRIPTION:
Patients with chronic kidney disease (CKD) develop anemia due to reduced erythropoietin production by the kidney. Correction of anemia has been shown to improve exercise capacity, cognition, quality of life and may slow disease progression.

The primary objective of this study is to compare the change in hemoglobin (Hb) that occurs from study start to the end of the study in pre-dialysis patients with anemia of chronic kidney disease (CKD) who are receiving PROCRIT (epoetin alfa) once every two weeks (Q2W) and once every four weeks (Q4W). This study will enroll 259 patients who will be randomly assigned (assigned to a treatment group by chance) to receive epoetin alfa subcutaneously (SC, under the skin) at one of four doses.

This study will have a Screening Phase of up to one week when patients will be evaluated for study eligibility followed by an open-label Treatment Phase of 16 weeks when patients will be randomly assigned to receive epoetin alfa administered under the skin at one of four dosing regimens. Patients will then complete a Post-Treatment Follow-Up Phase of 1 week (Week 17). Hemoglobin will be measured weekly. There will be no dose adjustments during the initial 4 weeks of the study, however, the dose may be withheld during this time if necessary. Further dose increases may occur at 4-week intervals and dose reductions may occur as frequently as the dosing interval assigned at randomization.

Patients will be eligible for epoetin alfa dose adjustments starting at the Week 5 visit if Hb is > 12 g/dL or Hb increases too rapidly (e.g., >1.0 g/dL in the last one or two consecutive weeks). The last dose of epoetin alfa administered for any treatment group will coincide with the dosing frequency assigned to that group. Epoetin alfa will not be administered later than Week 16 for any treatment group.

Hematology, serum chemistry, and iron status will be assessed at intervals throughout the study. The number of units of blood transfused, pre-transfusion Hb level, and the reasons for transfusion will be collected. Clinical laboratory results, vital signs, and the incidence and severity of adverse events will be assessed and monitored during the study.

Protocol Addendum: An Open-Label Extension of PROCRIT (Epoetin alfa) Maintenance Therapy Administered Every Six Weeks (Q6W) for the Treatment of Anemia of Chronic Kidney Disease (CKD). The Main Protocol, as described above, was designed to evaluate whether patients with anemia of CKD could be started on epoetin alfa therapy at one of four dosing regimens: 10,000 U once every week, 20,000 U every two weeks, 20,000 U every 4 weeks, or 40,000 U every four weeks. As an addendum to the Main Protocol, up to sixty (60) patients completing the original protocol with a hemoglobin (Hb) between 11 and 12 g/dL will be given an opportunity to enroll in an open-label extension study that will begin at the end of the Main Protocol timeline (Week 17). The primary objective of this open-label extension is to evaluate if epoetin alfa 40,000 U given SC every six weeks (Q6W), can maintain Hb within the range of 11-12 g/dL in patients with anemia of chronic kidney disease (CKD).

This open-label extension will have a Screening Phase of up to one week (during Week 17) when patients will be evaluated for eligibility, an Open-Label Treatment Phase of 12 weeks duration (Weeks 18-Week 30), and a Post-Treatment Follow-Up Phase of 6 weeks (ending at Week 36 or 6 weeks from the date of the last dose of epoetin alfa). All patients will receive a first dose of epoetin alfa 40,000 U SC every 6 weeks beginning with Week 18, a second dose at Week 24, and a third and final dose at Week 30. During the Treatment Phase, Hb will be measured weekly. Dosing will not be increased during the open-label extension. A six-week follow-up period is required after administration of the Week 30 dose for those patients receiving all 3 doses. If Hb falls below 10 g/dL at any time or if the patient requires a red blood cell (RBC) transfusion, the patient will be withdrawn from the open-label extension, and the Post-Treatment Follow-Up Phase will occur 6 weeks later.

Hematology, serum chemistry, and iron status will be assessed at intervals throughout the study. The number of units of blood transfused, pre-transfusion Hb level, and the reasons for transfusion will be collected. Clinical laboratory results, vital signs, and the incidence and severity of adverse events will be assessed and monitored during the study. Patients will receive epoetin alfa under the skin (SC) at a dose of 10,000 units (U) every week, 20,000 U every 2 weeks, 20,000 U every 4 weeks or 40,000 U every 4 weeks for 16 weeks. Protocol Addendum: Patients will receive epoetin alfa 40,000 U every 6 weeks over 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have CKD with Hg level <11 g/dL at study start
* must not have received any erythropoietic agents within 8 weeks of study start
* Patients with reproductive potential and their partners must practice an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, partner sterilization) before entry and throughout the study, female subjects with reproductive potential must have a negative urine pregnancy test within 7 days of the first dose of epoetin alfa
* Patients must have signed informed consent documents indicating that they agree to participate in the study, including the completion of all study-related procedures and evaluations.

Protocol Addendum: Patients must have participated in the Main Protocol of this study and completed all study-related procedures

* Patients must have a Hb between 11-12 g/dL at baseline (measured by HemoCue)
* Patients must have CKD defined as glomerular filtration rate (GFR) >=15 to <=90 mL/min as determined using the Modification of Diet for Renal Disease (MDRD) equation.

Exclusion Criteria:

* No patients receiving dialysis or scheduled to receive dialysis during the course of the study
* No patients with a current diagnosis of poorly controlled hypertension after adequate antihypertensive therapy or those with severe congestive heart failure (New York Heart Association Class IV), or known severe stable or unstable coronary artery disease
* No patients receiving chemotherapy for cancer within 3 months prior to study start or expected during study participation
* No patients with a current diagnosis of anemia due to Vitamin B12 deficiencies, hemolysis, or gastrointestinal bleeding or a history of/or active blood or bleeding disorders (this includes but is not limited to porphyria, thalassemia, myelodysplastic syndrome, and sickle cell anemia. No patients with liver diseases or any other diseases known to cause anemia
* No patients with a past history of thrombotic vascular events, (including but not limited to stroke, transient ischemic attack, myocardial infarction, coronary artery disease, and deep venous thrombosis) within the past 5 years
* No patients with a life expectancy of <= 6 months
* No women who are currently pregnant or lactating. No patients previously unresponsive to erythropoietic agents.

Protocol Addendum: No patients with a transferrin saturation (TSAT) <20% and a ferritin <50 ng/mL

* No patients with an epoetin alfa dose reduction/hold within the past four weeks of treatment in the Main Protocol, for a Hb rate of rise (>1 g/dL over 1 or 2 consecutive weeks),or a Hb above 12 g/dL
* No patients with iron overload defined as a TSAT > 70% or a ferritin > 1000 ng/mL
* No patients with a serum albumin concentration < 2.6 g/dL, or unstable angina
* No patients with chemotherapy for cancer within 3 months prior to baseline or expected during open-label extension participation
* No patients with known solid tumor malignancy or with new onset seizures within 3 months or seizures not controlled by medication prior to baseline. No patients receiving transfusion of platelets or packed red blood cells within 28 days prior to the first dose of epoetin alfa. No patients who have been previously unresponsive to erythropoietic agents, including patients who were treatment failures during the Main Protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2005-09; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin (Hb) from baseline to the end of the study; Primarily interested in the change in Hb between Q2W vs Q4W groups. Protocol Addendum: Hb change from baseline to end of open-label extension (no more than 36 weeks)

SECONDARY OUTCOMES:
Hb response (defined as achieving a Hb increase =>1g/dL from baseline any time during study); Change in Hb over time; Treatment failures; Blood transfused; Epoetin alfa dose when Hb is achieved and at study end.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Spinowitz B, Germain M, Benz R, Wolfson M, McGowan T, Tang KL, Kamin M; Epoetin Alfa Extended Dosing Study Group. A randomized study of extended dosing regimens for initiation of epoetin alfa treatment for anemia of chronic kidney disease. Clin J Am Soc Nephrol. 2008 Jul;3(4):1015-21. doi: 10.2215/CJN.05681207. Epub 2008 Apr 9. PMID 18400964
- See also: An Open-Label, Randomized, Multicenter Study of the Initiation of Four Dosing Regimens of PROCRIT (Epoetin alfa) for the Treatment of Anemia of Chronic Kidney Disease (CKD) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=526&filename=CR003397_CSR.pdf
- See also: An Open-Label, Randomized, Multicenter Study of the Initiation of Four Dosing Regimens of PROCRIT (Epoetin alfa) for the Treatment of Anemia of Chronic Kidney Disease (CKD) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=526&filename=CR003397_CSR2.pdf